CLINICAL TRIAL: NCT03867331
Title: A Phase I Dose Escalation Study With Controlled Human Malaria Infection (CHMI) to Assess the Safety, Immunogenicity and Efficacy of VLPM01 in Healthy, Malaria-Naïve Volunteers
Brief Title: To Assess the Safety, Immunogenicity and Efficacy of VLPM01 in Healthy, Malaria-Naïve Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VLP Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VLPM01-01 WRAIR #2568
Record Dates: First submitted 2019-02-28; First posted 2019-03-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 microgram VLPM01 (Experimental): 5 microgram doses of VLPM01 vaccine, intramuscular administration, n=10
  Interventions: Biological: 5 microgram VLPM01
- 15 microgram VLPM01 (Experimental): 15 microgram doses of VLPM01 vaccine, intramuscular administration, n=10
  Interventions: Biological: 15 microgram VLPM01
- 30 microgram VLPM01 (Experimental): 30 microgram doses of VLPM01 vaccine, intramuscular administration, n=10
  Interventions: Biological: 30 microgram VLPM01
- Controlled Human Malaria Infection (CHMI) Phase (Experimental): Infectivity Control Participants, n=6
  Interventions: Other: Plasmodium falciparum challenge

INTERVENTIONS:
Biological: 5 microgram VLPM01 — VLPM01 is an alpha-VLP pre-erythrocytic malaria vaccine which targets circumsporozoite protein (CSP), adjuvanted with 0.75 mg alum.
  Arms: 5 microgram VLPM01
Biological: 15 microgram VLPM01 — VLPM01 is an alpha-VLP pre-erythrocytic malaria vaccine which targets circumsporozoite protein (CSP), adjuvanted with 0.75 mg alum.
  Arms: 15 microgram VLPM01
Biological: 30 microgram VLPM01 — VLPM01 is an alpha-VLP pre-erythrocytic malaria vaccine which targets circumsporozoite protein (CSP), adjuvanted with 0.75 mg alum.
  Arms: 30 microgram VLPM01
Other: Plasmodium falciparum challenge — Expose forearms to five (5) Plasmodium falciparum (strain NF54; clone 3D7) bites
  Arms: Controlled Human Malaria Infection (CHMI) Phase

SUMMARY:
This study is a proof-of-concept, first in human, Phase I, single center study designed to evaluate the safety, tolerability, immunogenicity and experimental efficacy of VLPM01 in healthy, malaria-naïve adult volunteers. The VLPM01 product will be adjuvanted with alhydrogel. The study design was based on the FDA's guidance "General Principles for the Development of Vaccines to protect Against Global Infectious Diseases" (2011).

DETAILED DESCRIPTION:
The study will have four (4) phases: Screening, Dose Escalation, Controlled Human Malaria Infection (CHMI) and Follow-Up. The study will be conducted at the Walter Reed Army Institute of Research in Silver Spring, Maryland (WRAIR), as this institute has extensive experience in conducting clinical studies of malaria vaccines with CHMI.

A total of 36 participants will be enrolled in this study. Thirty (30) eligible participants will participate in the Dose Escalation Phase as vaccinees and 6 eligible participants will be added during the CHMI Phase to act as infectivity controls. Up to 6 additional eligible participants will serve as alternate vaccinees during the Dose Escalation Phase and up to 6 eligible participants will as act as alternate infectivity controls during the CHMI Phase. Alternates are only enrolled if a designated vaccinee is not eligible on the day of first vaccination or if a designated infectivity control is not eligible on the Day of Challenge. Withdrawn participants will not be replaced.

ELIGIBILITY:
Inclusion Criteria: It should say meet all the following criteria:

1. Healthy adults between the ages 18-49 (inclusive);
2. Able and willing to provide written, informed consent;
3. Able and willing to comply with all research requirements, in the opinion of the Investigator;
4. Agreement to refrain from blood donation during the course of the study. Volunteers who have undergone CHMI can donate to other research once the study is complete but cannot donate to the American Red Cross for at least three (3) years after the CHMI event;
5. Laboratory Criteria within 56 days before enrollment:

   * Hemoglobin ≥ 11.7 g/dL for women; ≥ 12.0 g/dL for men;
   * White Blood Cell count = 3,800-10,800 cells/mm3;
   * Platelets = 140,000-400,000/mm3;
   * Alanine aminotransferase (ALT; SGPT) 9-46 U/L male and 6-29 U/L female;
   * Serum creatinine ≤ 1.5 mg/dL;
   * Negative HIV testing (HIV Ab / antigen 4th generation screen with reflex confirmatory RNA testing);
   * Negative hepatitis B surface antigen (HBsAg) and hepatitis C antibody testing;
6. Birth control requirements:

   Female participants must meet one of the following two (2) criteria:
   * No reproductive potential due to post-menopausal status (12 months of natural [spontaneous] amenorrhea) or hysterectomy, bilateral oophorectomy or tubal ligation;
   * Women of childbearing potential should agree to practice highly effective contraception at least 30 days before enrollment and through 60 days post-CHMI or post-last vaccination (whichever is latest), using one of the following methods: condoms (male or female) with spermicide; diaphragm, or cervical cap with spermicide; intrauterine device; contraceptive pills, patch, injection, intravaginal ring or other FDA-approved contraceptive method; male partner has previously undergone a vasectomy; abstinence.

   Male participants are encouraged but not required to practice highly effective contraception to avoid pregnancy in their partner from 30 days prior to enrollment through 60 days post-CHMI.
7. For all female participants a negative β-HCG pregnancy test (urine) on day of enrollment, each day of vaccination, and the day of CHMI;
8. Reachable (24/7) by mobile phone during the period between CHMI and 28 days post-CHMI, per volunteer report;
9. No plans to travel outside the Washington DC metro area between the day of challenge and 28 days post-challenge;
10. If a participant is active duty military, he or she must obtain approval from his or her supervisor per WRAIR Policy 11-45;
11. Must have low (<10%) cardiac risk factors according to clinical Gaziano criteria assessed at screening, and a normal or normal variant ECG;
12. Completion of Study Comprehension Quiz (minimum passing score of 70% with 3 attempts permitted).

Exclusion Criteria: Should meet anyone of the following criteria:

1. History of malaria infection (any species) or residence in a malaria-endemic area for more than 5 years
2. History of serology-confirmed or suspected chikungunya virus (CHIKV) infection;
3. Previous travel to malaria endemic regions within the past three (3) months before study enrollment defined as first vaccination or day of challenge (for infectivity controls) or planned travel to malaria endemic regions during the vaccination, CHMI and follow-up period;
4. Any history of receiving a malaria vaccine or chikungunya vaccine;
5. Received an investigational product in the 30 days before enrollment, or planned to receive during the study period;
6. Participation in another clinical research study that would require excessive blood draws in conjunction with this study (as determined by the investigator)
7. Receipt of immunoglobulins or blood products within three (3) months before enrollment;
8. Any history of anaphylaxis;
9. History of sickle cell trait or disease, or any condition that could affect susceptibility to malaria infection, per patient verbal report;
10. Pregnancy, lactation or intention to become pregnant during the study;
11. Contraindications or allergies to the use of all three (3) proposed anti-malarial medications; Malarone (atovaquone/proguanil), Coartem (artemether/lumefantrine) and Chloroquine; contraindication to one or two is not exclusionary;
12. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ);
13. History of autoimmune disease;
14. Significant (e.g. systemic anaphylaxis) hypersensitivity reactions to mosquito bites (local reactions at the site of mosquito bites are not an exclusion criterion);
15. Suspected or known current alcohol or drug abuse as defined by an alcohol intake of greater than three (3) drinks a day on average for a man, and greater than two (2) drinks a day on average for a woman for a period of 12 months before enrollment;
16. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent;
17. Any clinically significant abnormal finding on chemistry or hematology blood tests or clinical examination, not already specified, as determined by the Investigator;
18. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data, in the opinion of the Investigator;
19. Current anti-tuberculosis prophylaxis or treatment;
20. History of splenectomy;
21. History of confirmed or suspected immunodeficiency;
22. Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema;
23. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two (2) years;
24. Diabetes mellitus (type I or II), with the exception of gestational diabetes;
25. Thyroid disease;
26. Idiopathic urticaria within the past year;
27. Hypertension that is not well controlled by medication or is more than 150/95 at enrollment;
28. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws;
29. Chronic or active neurologic disease to include seizure disorder and chronic migraine headaches. Exceptions are: i) childhood febrile seizures, or ii) seizures secondary to alcohol withdrawal more than three [3] years ago;
30. Participants receiving any of the following substances:

    * Systemic immunosuppressive medications or cytotoxic medications within 12 weeks before enrollment [with the exception of a short course of corticosteroids (≤14 days duration or a single injection) for a self-limited condition at least two (2) weeks before enrollment; inhaled, intranasal or topical steroids are not considered exclusionary];
    * History of receipt of malaria prophylaxis within eight (8) weeks of CHMI;
    * Live attenuated vaccines within 28 days before initial study vaccine administration;
    * Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, planned for administration seven (7) days before or after study vaccine administration;
31. History of arthritis diagnosis, either rheumatoid, osteoarthritis or any other type
32. History of other diagnosed rheumatoid disorders.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited local reactogenicity to VLPM01 at 5, 15 and 30 μg in the 7 days following vaccination | 7 days following vaccination
Occurrence of solicited systemic reactogenicity to VLPM01 at 5, 15 and 30 μg in the 7 days following vaccination | 7 days following vaccination
Occurrence of unsolicited adverse events related to VLPM01 at 5, 15 and 30 μg in the 7 days following vaccination | 7 days following vaccination
Occurrence of adverse events of special interest during follow-up period | through study completion, an average of 18 months
Number of participants experiencing any serious adverse event after vaccination. | through study completion, an average of 18 months

SECONDARY OUTCOMES:
Anti-CSP IgG levels measured by ELISA | day 113 after third dose
Positive thick blood smear test for P. falciparum malaria following CHMI | day 6 to day 20 post challenge
Time to first positive thick blood smear test for P. falciparum following CHMI | day 6 to day 20 post challenge
  Number of subjects with Plasmodium Falciparum parasitemia defined by a positive blood slide, following sporozoite challenge
Percentage of participants with a minimum threshold of >20 μg/ml anti-CSP IgG after vaccination as measured by ELISA. | day 15 to post day 113 after third dose

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Institute of Research, Bethesda, Maryland, United States